CLINICAL TRIAL: NCT06945588
Title: The Influence of Different Music Genres on Hearing Performance in Noise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Merve MERAL ÇETİNKAYA, Assist. Prof., Istanbul Aydın University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 09/990
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hearing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Happy music (Experimental)
  Interventions: Behavioral: Music listening
- Sad music (Experimental)
  Interventions: Behavioral: Music listening
- No music (No Intervention)

INTERVENTIONS:
Behavioral: Music listening — Happy music group listened to happy music (major mode with a tempo of >120 beats per minute).
  Arms: Happy music
Behavioral: Music listening — Sad music group listened to sad music (minor mode with a tempo of <80 beats per minute).
  Arms: Sad music

SUMMARY:
A fast tempo and major mode music improves cognitive performance by triggering a feeling of happiness. This study examines the impact of music on hearing performance, hypothesizing that listening to happy music may improve hearing performance in noise. Sixty-three normal hearing subjects aged between 18 and 35 years old were included. The subjects were randomly assigned to three groups: happy music, sad music, and control groups. The songs composed in minor mode with a tempo of <80 beats per minute were categorized as "sad," while songs composed in major mode with a tempo of >120 beats per minute were categorized as "happy". The Audible Contrast Threshold (ACT) Test and Hearing in Noise Test (HINT) were administered before and immediately after playing the music tracks. Repeated measures ANOVA test was run to compare the changes in measurement scores before and after listening to music.

ELIGIBILITY:
Inclusion Criteria:

* Native Turkish speakers,
* Aged between 18 and 35 years old with normal hearing thresholds (pure tone average <25 dB),
* No history of otologic, psychiatric, or neurologic diseases

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
The change in hearing performance in noise will be examined with Turkish Hearing in Noise Test after listening to different music genres. | Before and immediately after playing the music tracks.
  Turkish Hearing in Noise Test (HINT): The adaptive test protocol was followed through two JBL Control One loudspeakers. The chair was placed at a distance of one meter from the loudspeaker, at a 90° angle to each other and aligned with the participant's ear level in the horizontal plane, as described in the HINT protocol. The evaluation was performed in three conditions: noise front condition (speech and noise 0°), noise right condition (speech 0°, noise 90°), and noise left condition (speech 0°, noise 270°).

SECONDARY OUTCOMES:
The change in hearing performance in noise will be examined with Audible Contrast Thresholdafter listening to different music genres. | Before and immediately after playing the music tracks.
  Audible Contrast Threshold (ACT) Test: Some noise samples were Spectro temporally modulated (such as a siren sound). The patient was asked to press a button when they heard the siren sound (Zaar et al., 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No